CLINICAL TRIAL: NCT06859047
Title: Comprehensive Hemodynamic Assessment Via Echocardiography: the Echodynamic Approach Compared to Right Heart Catheterization
Brief Title: The Echodynamic Approach
Acronym: TECH
Status: Recruiting | Type: Observational
Sponsor: IRCCS Ospedale San Raffaele (Other)
Responsible Party: Principal Investigator, Carlo Gaspardone, Medical Doctor, IRCCS Ospedale San Raffaele
Other Study IDs: TECH-HSR-2025
Record Dates: First submitted 2025-02-22; First posted 2025-03-05 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Echocardiography, Transthoracic; Right-heart Hemodynamics
Keywords: hemodynamics; right heart catheterization; echocardiography; echodynamics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The aim of this prospective observational study is to assess the accuracy of non-invasive hemodynamic parameter estimation via trans-thoracic echocardiography (TTE) compared to the invasive gold standard of right heart catheterization (RHC). This study will include patients who undergo both TTE and RHC on the same day, under the same hemodynamic conditions. The primary research question is: how does the echodynamic evaluation perform compared to right heart catheterization?

DETAILED DESCRIPTION:
The non-invasive echocardiographic assessment will be used to esimate via mathematic formulas all the direct and indirect paramethers obtained from the right side catheterization. Each value obtained from the model using echocardiographic paramethers will be compared to the invasive finding.

ELIGIBILITY:
Inclusion Criteria:

* Clinical need for an invasive hemodynamic assessment and an echocardiographic evaluation on the same day

Exclusion Criteria:

* Incomplete hemodynamic assessment for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients from multiple centers who received, within a short time frame (the same day), an invasive assessment of hemodynamic parameters through right heart catheterization and a non-invasive assessment through echocardiography.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Cardiac output | Baseline
  The primary outcome will be to compare the estimated value using echocardiographic parameters with the same invasive measurement by right heart catheterization recorded on the same day to avoid different cardiac load conditions. Right heart catheterization will be from either femural or jugular vein approach. The measure's unit will be L/min and L/min/m^2 for the indexed value.
Pulmonary artery pressure | Baseline
  The primary outcome will be to compare the estimated values using echocardiographic parameters with the same invasive measurement by right heart catheterization recorded on the same day to avoid different cardiac load conditions. Right heart catheterization will be from either femural or jugular vein approach. The measure's unit will be in mmHg, and it will be expressed as systolic, mean and diastolic pulmonary pressure.
Pulmonary vascular resistance | Baseline
  The primary outcome will be to compare the estimated values using echocardiographic parameters with the same invasive measurement by right heart catheterization recorded on the same day to avoid different cardiac load conditions. Right heart catheterization will be from either femural or jugular vein approach. The measure's unit will be in Woods Units
Right atrial pressure | Baseline
  The primary outcome will be to compare the estimated values using echocardiographic parameters with the same invasive measurement by right heart catheterization recorded on the same day to avoid different cardiac load conditions. Right heart catheterization will be from either femural or jugular vein approach. The measure's unit will be in mmHg.

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - Ospedale Generale regionale "F.Miulli", Bari
  - IRCCS Ospedale San Raffaele, Milan
  - IRCCS Policlinico San Matteo Pavia, Pavia

IPD SHARING:
Plan to Share IPD: Undecided